CLINICAL TRIAL: NCT04771377
Title: Effect of Protein Supplementation and a Structured Physical Exercise Program on Changes in Body Composition, Metabolic Flexibility (Energy Consumption of Substrates), and Functionality in Women During Weight Loss Induced by BS
Brief Title: Effect of Protein Supplementation and a Structured Exercise Program on Muscle in Women After Bariatric Surgery.
Acronym: SarcoFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Garmin International (Industry); Institut Nacional d'Educacio Fisica de Catalunya (Other)
Responsible Party: Principal Investigator, Violeta Moizé, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2020/0028
Record Dates: First submitted 2021-02-11; First posted 2021-02-25 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenic Obesity; Bariatric Surgery Candidate; Nutritional Deficiency; Protein Intolerance
Keywords: Sarcopenia; Physical training; Postmenopausal Women
MeSH Terms: conditions — Malnutrition; Sarcopenia | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: 2:2:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard protein supplementation (SPS) (Experimental): 0.8g protein/ IBW/ day
  Interventions: Dietary Supplement: Protein Supplementation
- High protein supplementation (HPS) (Experimental): 1.2g protein/ IBW/ day
  Interventions: Dietary Supplement: Protein Supplementation
- HPS + PA (Experimental): 1.2g protein/ IBW/ day + PA 3 times a week/ 12 weeks
  Interventions: Dietary Supplement: Protein Supplementation

INTERVENTIONS:
Dietary Supplement: Protein Supplementation — protein supplements will be supplied to participants at no cost physical activity Will be performed virtually by PT
  Other Names: Physical training; standard protein supplementation

SUMMARY:
Obesity is considered a chronic disease that increases the risk of developing diseases that reduce life expectancy. The treatment of obesity is complex. However, treatments based exclusively on dietary changes have not shown long-term efficacy especially in people with severe obesity. In contrast, in this group of people bariatric surgery (BS) has shown good long-term results in weight loss and maintenance. These changes are accompanied by significant improvements in health, improved quality of life, and reduced mortality. However, the changes in the digestive system created by BS and the high level of dietary restriction, affect the nutritional status and require a proper supplementation of vitamins and minerals during the follow-up. Intense weight loss during the first few months, coupled with an insufficient amount of protein in the diet, can lead to a loss of muscle mass. Excessive muscle loss during the short-term period can lead to functional repercussions (decreased strength and physical function) and reduced calories that the body burns daily. Naturally, this is especially important in people suffering from sarcopenia before BS, and it occurs more frequently in postmenopausal women. Despite this is known, specific protein intake recommendations after BS have not yet been defined based on scientific evidence. In this context, the first part of our proposal will assess the effect of two levels of protein supplementation: standard (S-PS) versus high (H-PS) on changes in a) body composition, b) energy expenditure, c) metabolic flexibility d) the physical condition during weight loss that follows BS. In addition, in patients with H-PS, the added effect of a physical exercise program, carried out with a personal trainer (professional of sports medicine trainer) virtually, will be evaluated. Protein supplementation and the virtual exercise program will be done during the 4 months following BS, and the results will be studied at 4, 8, and 12 months. Once the results have been defined, it is essential to transfer the recommendations to the real world. In a second part, and to achieve knowledge transfer to clinical practice, the investigators will explore the key elements that influence patient experience (XPA).

DETAILED DESCRIPTION:
Obesity is considered a chronic disease that increases the risk of developing diseases that reduce life expectancy. The treatment of obesity is complex. However, treatments based exclusively on dietary changes have not shown long-term efficacy especially in people with severe obesity. In contrast, in this group of people bariatric surgery (BS) has shown good long-term results in weight loss and maintenance. These changes are accompanied by significant improvements in health, improved quality of life, and reduced mortality. However, the changes in the digestive system created by BS and the high level of dietary restriction, affect the nutritional status and require a proper supplementation of vitamins and minerals during the follow-up. Intense weight loss during the first few months, coupled with an insufficient amount of protein in the diet, can lead to a loss of muscle mass. Excessive muscle loss during the short-term period can lead to functional repercussions (decreased strength and physical function) and reduced calories that the body burns daily. Naturally, this is especially important in people suffering from sarcopenia before BS, and it occurs more frequently in postmenopausal women. Despite this is known, specific protein intake recommendations after BS have not yet been defined based on scientific evidence. In this context, the first part of our proposal will assess the effect of two levels of protein supplementation: standard (SP-S) versus high (SP-A) on changes in a) body composition, b) energy expenditure, c) metabolic flexibility d) the physical condition during weight loss that follows BS. In addition, in patients with SP-Alta, the added effect of a physical exercise program, carried out with a personal trainer (professional of sports medicine trainer) virtually, will be evaluated. Protein supplementation and the virtual exercise program will be done during the 4 months following CO, and the results will be studied at 4, 8, and 12 months. Once the results have been defined, it is essential to transfer the recommendations to the real world. In a second part, and to achieve knowledge transfer to clinical practice, the investigators will explore the key elements that influence patient experience (XPA). The investigators will define indicators to assess it, especially those that are related to adherence to nutritional recommendations and to changes in lifestyle. The investigators are currently in the recruitment phase of the study. I have studied the necessary elements, ambitions and included the components that will help to define the dietary and lifestyle recommendations for our population. Aim to facilitate and define the performance of the professionals providing realistic, based on the XPA and in this way to improve the impact of the CO on health and quality of life. This is an ambitious and necessary study and includes all the component that will help define dietary and lifestyle recommendations for our population. It aims to facilitate and define the action of professionals provides realistic tools, based on XPA and thus improve the impact of BS on health and quality of life.

Description of the population to study sedentary women, candidates for BS at our institution.

ELIGIBILITY:
Inclusion Criteria:

women ≥45 years of age who meet CB criteria: Body mass index (BMI) ≥40.0 kg / m2 or between 35.0 and 39.9 kg / m2 with comorbidities (metabolic diseases, cardiorespiratory diseases), sedentary lack of regular physical activity: <30 minutes / day and <3 days / week).

Exclusion Criteria:

* presence of severe joint disease, severe liver disease, history of cardiovascular event or known heart disease, renal failure (defined as a FG <30 ml / min), type 1 or type 2 diabetes with HbA1c> 10%, being treated with drugs that may affect body composition (such as corticosteroids), exercise muscle strength-endurance regularly (more than 2 times / week), have previously undergone obesity surgery.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will only include women. The difference in muscle mass and strength justifies the need for this limitation. In addition, women account for 80% of CB cases in our Hospital and in the vast majority of literature series. Given that muscle mass loss and risk of sarcopenia are typical of older adults, our study (focused on the prevention and / or delay of the onset of sarcopenia) targets women over the age of 45 a first CB in our center. Although the results of this study will only be valid for this group, the resulting nutritional and lifestyle recommendations will be relevant as women are the majority in the use of CB. Addressing this goal in men would require a different protocol.
Enrollment: 75 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
effect of PS and PA on Changes in fat mass and Fat free mass (kg) | 4 months after BS
  change from baseline in DEXA values
effect of PS and PA on Changes in fat mass and Fat free mass (kg) | 8 months after BS
  change from baseline in DEXA values
effect of PS and PA on Changes in fat mass and Fat free mass (kg) | 12 months after BS
  change from baseline in DEXA values
effect of PS and PA on resting energy expenditure (REE) (Kcal/ day) | 4 months after BS
  change from baseline in estimated REE from indirect calorimety
effect of PS and PA on resting energy expenditure (REE) (Kcal/ day) | 8 months after BS
  change from baseline in estimated REE from indirect calorimety
effect of PS and PA on resting energy expenditure (REE) (Kcal/ day) | 12 months after BS
  change from baseline in estimated REE from indirect calorimety
Strength | 4 months after BS
  changes from baseline on prediction of ne repetition máximum (1-RM) and hang grip.
Strength | 8 months after BS
  changes from baseline on prediction of ne repetition máximum (1-RM) and hang grip.
Strength | 12 months after BS
  changes from baseline on prediction of ne repetition máximum (1-RM) and hang grip.
Functionality | 4 months after BS
  changes from baseline on sit and stand
Functionality | 8 months after BS
  changes from baseline on sit and stand
Functionality | 12 months after BS
  changes from baseline on sit and stand
Metabolic flexibility - oxidation of substrates: VO2 peak | 4 months after BS
  change in VO2 peak measured by Ergocard during half-effort test
Metabolic flexibility - oxidation of substrates: VO2 peak | 8 months after BS
  change in VO2 peak measured by Ergocard
Metabolic flexibility - oxidation of substrates: VO2 peak | 12 months after BS
  change in VO2 peak measured by Ergocard during half-effort test
Respiratory quotient | 4 months after BS
  change in RQ determined by Ergocard during half-effort test
Respiratory quotient | 8 months after BS
  change in RQ determined by Ergocard during half-effort test
Respiratory quotient | 12 months after BS
  change in RQ determined by Ergocard during half-effort test
Fat oxidation (FatMax) during during half-effort test | 4 months after BS
  Time to spend to reach the cross over pony for RQ=1 determined by Ergocard during half-effort test (min)
Fat oxidation (FatMax) during during half-effort test | 8 months after BS
  Time to spend to reach the cross over pony for RQ=1 determined by Ergocard during half-effort test (min)
Fat oxidation (FatMax) during during half-effort test | 12 months after BS
  Time to spend to reach the cross over pony for RQ=1 determined by Ergocard during half-effort test (min)
Adherence to PS (BCAA biomarker) | 4 months after BS
  serum change in BCAA (mcg)
Adherence to PS (BCAA biomarker) | 8 months after BS
  serum change in BCAA (mcg)
Adherence to PS (BCAA biomarker) | 12 months after BS
  serum change in BCAA (mcg)
Adherence to PS (urinary nitrogen 24hs.) | 4 months after BS
  Nitrogen (mg) values quantified in 24hs urine
Adherence to PS (urinary nitrogen 24hs.) | 8 months after BS
  Nitrogen (mg) values quantified in 24hs urine
Adherence to PS (urinary nitrogen 24hs.) | 12 months after BS
  Nitrogen (mg) values quantified in 24hs urine
Understand patients' priorities and the "painful points" of the care process. Explore the magnitude of these "painful points." This should make it possible to prioritize the areas to be evaluated. Test assessment tools | 12 months after BS
  identify by focus group patient reported outcomes by cualitative study

SECONDARY OUTCOMES:
Changes in BMI | 4 months after BS
  weight and height will be combined to report BMI in kg/m^2
Changes in BMI | 8 months after BS
  weight and height will be combined to report BMI in kg/m^2
Changes in BMI | 12 months after BS
  weight and height will be combined to report BMI in kg/m^2
Insulin sensitivity (HOMA-IR) | 4 months after BS
  fasting glucose (mg) and insulin (miliunits/ liter) will be combined to report Insulin sensitivity in
Insulin sensitivity (HOMA-IR) | 8 months after BS
  fasting glucose (mg) and insulin (miliunits/ liter) will be combined to report Insulin sensitivity in
Insulin sensitivity (HOMA-IR) | 12 months after BS
  fasting glucose (mg) and insulin (miliunits/ liter) will be combined to report Insulin sensitivity in

CONTACTS AND LOCATIONS:
Overall Officials: Violeta L Moizé, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No